CLINICAL TRIAL: NCT06729736
Title: Implementation of the Early Recovery After Surgery (ERAS) Protocol in Colorectal Cancer Patients: a Phase II Multi-Center, Prospective Single Arm Study
Brief Title: Implementation of the ERAS in Colorectal Cancer Patients: a Single Arm Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2410-124-1579
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: ERAS; Enhanced recovery; Early recovery; Colorectal surgery; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ERAS implemented arm (Experimental): ERAS protocol implemented patients (single arm).
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — The ERAS protocol includes:
  * Pre-admission education, counselling and nutritional support
  * Pre-induction oral analgesics
  * Minimal fasting and carbohydrate loading
  * Omission of nasogastric intubation
  * Intra-operative abdominal nerve block
  * Early mobilization
  * Early oral nutrition and minimal IV fluids
  * Multimodal opioid sparing analgesia
  * Postoperative nausea and vomiting prophylaxis
  * Early removal of urinary catheters

SUMMARY:
The goal of this study is to implement and investigate the efficacy of an Early Recovery After Surgery (ERAS) protocol in South Korean colorectal cancer patients.

The primary outcome will be the postoperative time taken to achieve the 'discharge criteria'.

Secondary outcomes will include adherence, hospital stay, early complications, mortality, pain scores, re-admission and quality of life questionnaire scores.

As a single arm study, all participants will be treated according to an ERAS protocol, which includes components such as early ambulation, minimal fasting, multimodal pain control and omission of- or early removal of invasive catheters.

DETAILED DESCRIPTION:
This multi-center prospective single arm clinical trial aims to investigate each component and item in the ERAS protocol implemented to perioperative care of colorectal cancer patients.

The primary endpoint will be the 'postoperative time to discharge criteria'. Discharge criteria will be defined as meeting all the criteria below:

* No fever
* Eating more than half of given solid diet
* No nausea or vomiting
* Gas passing or defecation
* Able to walk (more than 1 hour a day)
* No sign of surgical site infection
* Adequate pain control with oral analgesics such as acetaminophen and NSAIDs
* No sign of any other complication

Secondary outcomes will include:

* adherence of each ERAS item within the protocol
* postoperative hospital stay
* early postoperative complications (within 30 days of surgery)
* postoperative mortality
* postoperative pain scores (VAS scores)
* re-admission within 30 days of surgery
* Quality of Recovery questionnaire
* Health-related quality of life questionnaire

The specific ERAS protocol to be used in this study has been developed by Seoul National University Hospital, benchmarking the 2018 ERAS® society guidelines for colorectal surgery. The implementation process has been helped and guided by the ERAS® Implementation Program of the Encare team.

The ERAS protocol includes:

* Pre-admission education, counselling and nutritional support
* Pre-induction oral analgesics
* Minimal fasting and carbohydrate loading
* Omission of nasogastric intubation
* Intra-operative abdominal nerve block
* Early mobilization
* Early oral nutrition and minimal IV fluids
* Multimodal opioid sparing analgesia
* Postoperative nausea and vomiting prophylaxis
* Early removal of urinary catheters

This study aims to establish evidence on the factors affecting adherence and efficacy of each ERAS category, to guide a future pivotal RCT that will aim to develop a personalized, risk-stratified ERAS protocol that considers surgical risk and patient factors.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 19 years
* Pathologic diagnosis of colon cancer or rectal cancer
* Scheduled for minimally invasive (laparoscopic or robotic) colorectal cancer surgery
* Agreed to participate after a detailed explanation of the study

Exclusion Criteria:

* Stage 4 (distant metastasis)
* Emergency surgery
* Scheduled for transanal surgery
* Perforated colorectal cancer
* Obstructed colorectal cancer
* Familial colorectal cancer (HNPCC, FAP, MUYH polyposis, Peutz-Jeghers syndrome)
* Previous treatment for colorectal cancer
* History of other cancer within 5 years (excluding skin cancer)
* Acute infection
* Unable to read or understand the study
* Mental impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative time to discharge criteria | From the date of surgery until the date of first achieving all of the discharge criteria, assessed up to 100 days
  The time (days) from initiation of surgery to achieving the discharge criteria. Discharge criteria is defined as meeting all of the following criteria:
  * No fever
  * Eating more than half of given solid diet
  * No nausea or vomiting
  * Gas passing or defecation
  * Able to walk (more than 1 hour a day)
  * No sign of surgical site infection
  * Adequate pain control with oral analgesics such as acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDs)
  * No sign of any other complication

SECONDARY OUTCOMES:
Adherence to the ERAS protocol | From date of enrollment to the date of discharge after surgery, assessed up to 100 days
  Adherence to each item in the ERAS protocol
Hospital stay | From the date of hospital admission until the date of discharge after surgery, assessed up to 100 days
  Total length of hospital stay for surgery.
Early postoperative complication | From the day of surgery to the 30th postoperative day
  Postoperative complication within 30 days of surgery.
Postoperative mortality | From day of surgery until the end of clinical data gathering, assessed upto 100 days.
  Death caused by the surgery itself or any complication related to surgery.
Postoperative pain score: the Numeric Rating Scale (NRS) | From day of surgery until the end of clinical data gathering, assessed upto 100 days.
  Postoperative pain, evaluated using the Numeric Rating Scale (NRS) scale. This scale ranges from 0 to 10, with increasing values representing more severe pain.
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-10: Severe pain
  Pain scores at rest, and pain scores at movement will be collected and analyzed separately.
Re-admission within 30 days | From randomization until the end of clinical data gathering, assessed upto 100 days.
  Re-admission due to surgery complication within 30 days of surgery.
Health-related Quality of Life | From randomization until the end of clinical data gathering, assessed upto 100 days.
  Health related quality of life, assessed using the 5-level EQ-5D version (EQ-5D-5L) questionnaire.
  The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yong Jeong, M.D., Ph.D., Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No